CLINICAL TRIAL: NCT00656942
Title: Pain Responses in Patients on Long-Term Opioid Therapy for Chronic Pain
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jianren Mao, MD, PhD, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2003P 000110; MGH Fund # 1200-204727
Record Dates: First submitted 2008-04-09; First posted 2008-04-14 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Chronic Pain
Keywords: Pain
MeSH Terms: conditions — Chronic Pain; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Healthy: * subjects with no pain and no opioid treatment for at least six months
  * subjects receive quantitative sensory testing (QST)
  Interventions: Device: Quantitative Sensory Testing (QST)
- Pain, no opioid: * subjects have chronic pain but have not taken any opioid medication for at least 3 months
  * subjects receive QST
  Interventions: Device: Quantitative Sensory Testing (QST)
- Pain, opioid: * subjects have chronic pain and have been taking opioid medication for at least 3 months
  * subjects receive QST
  Interventions: Device: Quantitative Sensory Testing (QST)

INTERVENTIONS:
Device: Quantitative Sensory Testing (QST) — QST consists of a series of heat and cold stimulation tests.

SUMMARY:
The MGH Center for Translational Pain Research is seeking patients with chronic pain for a research study. The study is looking at the effect of opioid (narcotic) pain medicines on pain sensation, threshold and tolerance.

DETAILED DESCRIPTION:
The study consists of one visit, in which an interview, physical exam, lab work (urine test) and sensory testing will be done. The testing (Quantitative Sensory Testing) is noninvasive (no needles) and involves heat and cold stimulation. Compensation and some parking reimbursement provided.

ELIGIBILITY:
a. Inclusion/exclusion criteria

Inclusion Criteria for the group with chronic pain on chronic treatment with opioids:

1. Subject has chronic pain and is on stable chronic opioid treatment (morphine, fentanyl, oxycodone, methadone, hydromorphone, hydrocodone) for chronic pain for at least one month. We consider stable treatment if no change in the type and amount of daily opioid treatment for one month. Only patients with minimal daily opioid dose of at least 30 mg morphine equianalgesic dose will be included.
2. Subject is age 18 to 65 years.

Inclusion Criteria for the group with chronic pain on chronic treatment with non-opioids (currently not recruiting):

1. Subject has pain and is on stable chronic non-opioid treatment for chronic pain for at least one month.
2. Subject is age 18 to 65 years.

Inclusion Criteria for the group of opioid-naive healthy volunteers without chronic pain (currently not recruiting):

1. Subject is opioid naive meaning he/she did not receive chronic opioid treatment in the past or present, and did not receive acute treatment with opioids in the last 1 month
2. Subject does not have pain
3. Subject is age 18 to 65 years.

Exclusion Criteria for all groups:

1. Subject has lost tactile sensation in the sites for QST testing (upper extremities)
2. Subject has scar tissue or acute injury in the skin areas for QST testing (upper extremities)
3. Subject has neurological disease or a medical condition causing peripheral polyneuropathy and sensory changes (including but not limited to diabetes, alcoholism, AIDS, thyroid disease, liver or kidney disorders). It is the presence of neuropathy, not the causative disease itself, that is the exclusion criteria.
4. Subject had recent therapy that may influence QST results, e.g., neuroablative procedure involving upper extremities within six-months; peripheral neurolytic block within two-months; injection therapy for pain within four-weeks; sympathetic block within six months.
5. Subject has litigation pending relative to their chronic pain.
6. Subject has major psychiatric disorder (major depression disorder; bipolar disorder; schizophrenia; anxiety disorder; psychotic disorders; eating disorders; alcohol or drug dependence; attention deficit hyperactivity disorder); any known history of these conditions will exclude participation.
7. Subject has used illicit drugs within past 6 months.
8. Subject is pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The groups of subjects on chronic opioid and non-opioid treatment for chronic pain will be recruited from the MGH Pain Center's patients. We want to emphasize that our MGH Pain Center patient population comprehends a significant number of patients on stable dose of non-opioid and opioid pain medication for chronic pain. The investigators and study staff will search daily the MGH Pain Center clinic list and will approach the patients who might qualify for the study. The group of opioid naive subjects will be recruited by advertising in local newspapers and by using e-mail announcements through Partners HealthCare system.
Sampling Method: Non-Probability Sample
Enrollment: 419 (Actual)
Dates: Start 2006-07; Primary Completion 2013-10 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Response to warm/cold temperature | 2 hours
  Responses to warm/cold temperatures will be recorded by the Quantitative Sensory Testing device (QST).

CONTACTS AND LOCATIONS:
Overall Officials: Jianren Mao, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH Center for Translational Pain Center, Boston, Massachusetts, United States